CLINICAL TRIAL: NCT03697213
Title: An Online International Comparison of Thresholds for Triggering a Negative Response to the "Surprise Question"
Brief Title: The Surprise Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Radboud University Medical Center (Other); University of Bern (Other); Imperial College London (Other); Universiteit Antwerpen (Other); University of Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0253
Record Dates: First submitted 2018-09-25; First posted 2018-10-05 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Palliative Care; Terminal Illness
Keywords: Surprise Question; Prognostication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Practitioners: Registered General Practitioners in one of the six participating countries.
  Interventions: Other: Online study

INTERVENTIONS:
Other: Online study — 20 hypothetical patient summaries

SUMMARY:
This study investigates the use of the Surprise Question [SQ] (would you be surprised if this patient were to die in the next 12 months?) in routine practice. In particular, the study will investigate the consistency of the responses to the SQ and the relationship with the subsequent course of action decided upon.

DETAILED DESCRIPTION:
Whilst the original use of the Surprise Question was to identify people who might be in the last year of life and benefit from palliative care, the prognostic capability of the Surprise Question has been shown to be variable. What is unclear, is the extent to which a doctor should be "surprised" before a patient is suitable for palliative care, how consistently doctors respond to this question, and how the subsequent treatment decision relates to the SQ response.

The study will recruit 600 General Practitioners (GPs) from 6 participating countries (100 per country; UK, Germany, Switzerland, Italy, Belgium, the Netherlands). Each participant will asked to complete a series of 20 hypothetical patient summaries in an online task.

ELIGIBILITY:
Inclusion Criteria:

* Registered General Practitioner in one of the six participating countries
* Able to read and understand the language in which the questionnaire is presented to them

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of registered General Practitioners (GPs) with a variety of years of experience and seniority across six European countries will be approached to participate
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Probability estimate | Participants will have up to 8 months (until the study closes) to provide an estimate for each vignette (n=20)
  The continuous estimate of probability of dying within the next 12 months for the SQ (0-100%).

SECONDARY OUTCOMES:
The Surprise Question | up to 8 months (until the study closes)Participants will have up to 8 months (until the study closes) to provide a response for each vignette (n=20)
  Dichotomous response to the SQ (Yes/No)
The alternative Surprise Question | up to 8 months (until the study closes)Participants will have up to 8 months (until the study closes) to provide a response for each vignette (n=20)
  Dichotomous response to the alternative SQ (Yes/No)
Treatment options | up to 8 months (until the study closes)Participants will have up to 8 months (until the study closes) to provide a response for each vignette (n=20)
  The options for the course of action selected by the participants in each vignette

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, MA, MD, FRCP, Principal Investigator — University College, London
Locations (6):
- University of Antwerp, Antwerp, Belgium
- University of Mainz, Mainz, Germany
- University of Bologna, Bologna, Italy
- Radboud University Medical Centre, Nijmegen, Netherlands
- University Hospital of Bern, Bern, Switzerland
- Marie Curie Palliative Care Research Department, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] White N, Oostendorp LJ, Vickerstaff V, Gerlach C, Engels Y, Maessen M, Tomlinson C, Wens J, Leysen B, Biasco G, Zambrano S, Eychmuller S, Avgerinou C, Chattat R, Ottoboni G, Veldhoven C, Stone P. An online international comparison of palliative care identification in primary care using the Surprise Question. Palliat Med. 2022 Jan;36(1):142-151. doi: 10.1177/02692163211048340. Epub 2021 Oct 1. PMID 34596445
- [Derived] White N, Oostendorp L, Vickerstaff V, Gerlach C, Engels Y, Maessen M, Tomlinson C, Wens J, Leysen B, Biasco G, Zambrano S, Eychmuller S, Avgerinou C, Chattat R, Ottoboni G, Veldhoven C, Stone P. An online international comparison of thresholds for triggering a negative response to the "Surprise Question": a study protocol. BMC Palliat Care. 2019 Apr 9;18(1):36. doi: 10.1186/s12904-019-0413-x. PMID 30979361
- See also: The Study Protocol — https://bmcpalliatcare.biomedcentral.com/articles/10.1186/s12904-019-0413-x

DOCUMENTS (1):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT03697213/Prot_000.pdf